CLINICAL TRIAL: NCT00268216
Title: A Multicentre, Randomised, Double-blind, Parallel Group, Placebo-controlled Study to Investigate the Long-term Effects of Salmeterol/Fluticasone Propionate (Seretide tm) 50/500mcg BD, Salmeterol 50mcg BD and Fluticasone Propionate 500mcg BD, All Delivered Via the Diskus tm/Accuhaler tm Inhaler, on Mortality and Morbidity of Subjects With Chronic Obstructive Pulmonary Disease (COPD) Over 3 Years of Treatment
Brief Title: Survival Of Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCO30003
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: mortality; TORCH; SERETIDE; ADVAIR; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate; Fluticasone

INTERVENTIONS:
Drug: Salmeterol 50mcg/ Fluticasone Propionate 500mcg

SUMMARY:
The purpose of this study is to see if fluticasone 500mcg/salmeterol 50mcg can improve the survival of subjects with COPD and also assess the long term safety profile of this drug.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, parallel group, placebo controlled study to investigate the effects of salmeterol/fluticasone 50/500mcg bd, salmeterol 50mcg bd, and fluticasone 500mcg bd, all delivered via the DISKUS/ACCUHALER inhaler, on the survival of subjects with chronic obstructive pulmonary disease over 3 years of treatment.

ELIGIBILITY:
Inclusion criteria:

* Patients with COPD and FEV1 <60% of predicted normal and baseline (pre-bronchodilator) FEV1/FVC ratio <70%.
* Current or ex-smokers with a smoking history of at least 10 pack-years.

Exclusion criteria:

* Diagnosis of other respiratory disorders (including asthma).
* Requirement for long term oxygen therapy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6228 (Actual)
Dates: Start 2000-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
All cause mortality at 3 years

SECONDARY OUTCOMES:
Rate of moderate and severe COPD exacerbations and health status assessed by the St. George's Respiratory Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (385):
- United States (155):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Ozark, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Berkeley, California
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Luis Obispo, California
  - GSK Investigational Site, Sepuldeva, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Sunnyvale, California
  - GSK Investigational Site, Sylmar, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Arvada, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Loveland, Colorado
  - GSK Investigational Site, Pueblo, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Atlantis, Florida
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Longwood, Florida
  - GSK Investigational Site, Loxahatchee Groves, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pace, Florida
  - GSK Investigational Site, Palm Springs, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Zephyrhills, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Rome, Georgia
  - GSK Investigational Site, Roswell, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Champaign, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Hines, Illinois
  - GSK Investigational Site, North Chicago, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Swansea, Massachusetts
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, Livonia, Michigan
  - GSK Investigational Site, Saint Joseph, Michigan
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Gilford, New Hampshire
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, East Orange, New Jersey
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Trenton, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Bronxville, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Franklin, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Doylestown, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Ridley Park, Pennsylvania
  - GSK Investigational Site, Cranston, Rhode Island
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Milan, Tennessee
  - GSK Investigational Site, Morristown, Tennessee
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Chesapeake, Virginia
  - GSK Investigational Site, Fredericksburg, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Charleston, West Virginia
  - GSK Investigational Site, Huntington, West Virginia
  - GSK Investigational Site, La Crosse, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin
- Argentina (3):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Vicente López, Buenos Aires
- Australia (10):
  - GSK Investigational Site, Bankstown, New South Wales
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, North Gosford, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Toorak Gardens, South Australia
  - GSK Investigational Site, Frankston, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Austria (2):
  - GSK Investigational Site, Vienna
  - GSK Investigational Site, Wels
- Belgium (5):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Namur
  - GSK Investigational Site, Orp-Jauche
  - GSK Investigational Site, Ostend
  - GSK Investigational Site, Veurne
- Brazil (4):
  - GSK Investigational Site, Rio de Janeiro, Rio de Janeiro
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Santo André, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
- Bulgaria (4):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (14):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Maple Ridge, British Columbia
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Scarborough Village, Ontario
  - GSK Investigational Site, Thunder Bay, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Chile (3):
  - GSK Investigational Site, Temuco, Región de La Araucania
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- China (8):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wangfujing, Beijing
- GSK Investigational Site, Zagreb, Croatia
- Czechia (5):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Jaroměř
  - GSK Investigational Site, Ostrava - Fifejdy
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Tábor
- Denmark (4):
  - GSK Investigational Site, Aarhus C
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, København NV
  - GSK Investigational Site, Silkenborg
- Estonia (3):
  - GSK Investigational Site, Kohtal-Jdrve
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (8):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kinkomaa
  - GSK Investigational Site, Lappeenranta
  - GSK Investigational Site, Lohja
  - GSK Investigational Site, Mikkeli
  - GSK Investigational Site, Oulainen
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Vantaa
- France (23):
  - GSK Investigational Site, Annonay
  - GSK Investigational Site, Avrillé
  - GSK Investigational Site, Béthune
  - GSK Investigational Site, Bois-Guillaume
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Chamalières
  - GSK Investigational Site, Cholet
  - GSK Investigational Site, Corbeil Essonne
  - GSK Investigational Site, Férolles-Attilly
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lomme
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Maurepas
  - GSK Investigational Site, Meaux
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Quentin
  - GSK Investigational Site, Tarbes
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Verdun
- Germany (7):
  - GSK Investigational Site, Schwetzingen, Baden-Wurttemberg
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Greece (10):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Chania, Crete
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Kavala
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Maroussi, Athens
  - GSK Investigational Site, N. Efkarpia, Thessaloniki
  - GSK Investigational Site, Papagos/Athens
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Thessaloniki
- Hong Kong (5):
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, Kowloon
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Lai Chi Kok
  - GSK Investigational Site, Tai Po
- Hungary (6):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Cegléd
  - GSK Investigational Site, Dunaújváros
  - GSK Investigational Site, Szolnok
  - GSK Investigational Site, Tatabánya
  - GSK Investigational Site, Törökbálint
- Iceland (2):
  - GSK Investigational Site, Fossvogur. Reykjavic
  - GSK Investigational Site, Reykjavik
- Italy (7):
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Sesto San Giovanni (MI), Lombardy
  - GSK Investigational Site, Tradate (VA), Lombardy
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Bussolengo (VR), Veneto
- GSK Investigational Site, Riga, Latvia
- GSK Investigational Site, Kaunas, Lithuania
- Malaysia (4):
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kubang Kerian
  - GSK Investigational Site, Kuching
  - GSK Investigational Site, Tanjong Bungah
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- Netherlands (12):
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Bilthoven
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Dordrecht
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hoofddorp
  - GSK Investigational Site, Roosendaal
  - GSK Investigational Site, Terneuzen
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Zwolle
- New Zealand (5):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Wellington
  - GSK Investigational Site, Wellington South
- Norway (11):
  - GSK Investigational Site, Ålesund
  - GSK Investigational Site, Bardufoss
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Bodø
  - GSK Investigational Site, Harstad
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Sandvika
  - GSK Investigational Site, Skien
  - GSK Investigational Site, Trondheim
  - GSK Investigational Site, Tønsberg
  - GSK Investigational Site, Volda
- GSK Investigational Site, Lahore, Pakistan
- Philippines (3):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- Poland (5):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zabrze
- GSK Investigational Site, Ponce, Puerto Rico, Puerto Rico
- Romania (3):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
- GSK Investigational Site, Moscow, Russia
- GSK Investigational Site, Singapore, Singapore
- Slovakia (4):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Kráľovský Chlmec
  - GSK Investigational Site, Nové Zámky
  - GSK Investigational Site, Partizánske
- South Africa (4):
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Pretoria
- Spain (14):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Cartagena
  - GSK Investigational Site, Elda
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Orihuela/Alicante
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo/Pontevedra
  - GSK Investigational Site, Vizcaya
- Sweden (6):
  - GSK Investigational Site, Boden
  - GSK Investigational Site, Eksjö
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Helsingborg
  - GSK Investigational Site, Lidköping
  - GSK Investigational Site, Trollhättan
- Taiwan (5):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tau-Yuan County
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- GSK Investigational Site, Kiev, Ukraine
- United Kingdom (7):
  - GSK Investigational Site, Exeter, Devon
  - GSK Investigational Site, Bristol, Gloucestershire
  - GSK Investigational Site, Liverpool, Lancashire
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Newcastle upon Tyne, Northumberland
  - GSK Investigational Site, Headington, Oxfordshire
  - GSK Investigational Site, London
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Briggs AH, Glick HA, Lozano-Ortega G, Spencer M, Calverley PM, Jones PW, Vestbo J; TOwards a Revolution in COPD Health (TORCH) investigators. Is treatment with ICS and LABA cost-effective for COPD? Multinational economic analysis of the TORCH study. Eur Respir J. 2010 Mar;35(3):532-9. doi: 10.1183/09031936.00153108. Epub 2009 Aug 28. PMID 19717476
- [Background] Calverley PM, Anderson JA, Celli B, Ferguson GT, Jenkins C, Jones PW, Yates JC, Vestbo J; TORCH investigators. Salmeterol and fluticasone propionate and survival in chronic obstructive pulmonary disease. N Engl J Med. 2007 Feb 22;356(8):775-89. doi: 10.1056/NEJMoa063070. PMID 17314337
- [Background] Celli BR, Thomas NE, Anderson JA, Ferguson GT, Jenkins CR, Jones PW, Vestbo J, Knobil K, Yates JC, Calverley PM. Effect of pharmacotherapy on rate of decline of lung function in chronic obstructive pulmonary disease: results from the TORCH study. Am J Respir Crit Care Med. 2008 Aug 15;178(4):332-8. doi: 10.1164/rccm.200712-1869OC. Epub 2008 May 29. PMID 18511702
- [Background] Jenkins CR, Jones PW, Calverley PM, Celli B, Anderson JA, Ferguson GT, Yates JC, Willits LR, Vestbo J. Efficacy of salmeterol/fluticasone propionate by GOLD stage of chronic obstructive pulmonary disease: analysis from the randomised, placebo-controlled TORCH study. Respir Res. 2009 Jun 30;10(1):59. doi: 10.1186/1465-9921-10-59. PMID 19566934
- [Background] Crim C, Calverley PM, Anderson JA, Celli B, Ferguson GT, Jenkins C, Jones PW, Willits LR, Yates JC, Vestbo J. Pneumonia risk in COPD patients receiving inhaled corticosteroids alone or in combination: TORCH study results. Eur Respir J. 2009 Sep;34(3):641-7. doi: 10.1183/09031936.00193908. Epub 2009 May 14. PMID 19443528
- [Background] Ernst P, Suissa S. Pneumonia in elderly patients with chronic obstructive pulmonary disease. Curr Infect Dis Rep. 2008 May;10(3):223-8. doi: 10.1007/s11908-008-0037-4. PMID 18510885
- [Background] Ferguson GT, Calverley PMA, Anderson JA, Jenkins CR, Jones PW, Willits LR, Yates JC, Vestbo J, Celli B. Prevalence and progression of osteoporosis in patients with COPD: results from the TOwards a Revolution in COPD Health study. Chest. 2009 Dec;136(6):1456-1465. doi: 10.1378/chest.08-3016. Epub 2009 Jul 6. PMID 19581353
- [Background] Hanania NA. The impact of inhaled corticosteroid and long-acting beta-agonist combination therapy on outcomes in COPD. Pulm Pharmacol Ther. 2008;21(3):540-50. doi: 10.1016/j.pupt.2007.12.004. Epub 2008 Jan 6. PMID 18280761
- [Background] Houghton CM, Lawson N, Borrill ZL, Wixon CL, Yoxall S, Langley SJ, Woodcock A, Singh D. Comparison of the effects of salmeterol/fluticasone propionate with fluticasone propionate on airway physiology in adults with mild persistent asthma. Respir Res. 2007 Jul 14;8(1):52. doi: 10.1186/1465-9921-8-52. PMID 17629923
- [Background] Johnson M, Agusti AG, Barnes NC. Reflections on TORCH: potential mechanisms for the survival benefit of salmeterol/fluticasone propionate in COPD patients. COPD. 2008 Dec;5(6):369-75. doi: 10.1080/15412550802522924. PMID 19353351
- [Background] Keene ON, Vestbo J, Anderson JA, Calverley PM, Celli B, Ferguson GT, Jenkins C, Jones PW. Methods for therapeutic trials in COPD: lessons from the TORCH trial. Eur Respir J. 2009 Nov;34(5):1018-23. doi: 10.1183/09031936.00122608. PMID 19880616
- [Background] Drummond MB, Wise RA, John M, Zvarich MT, McGarvey LP. Accuracy of death certificates in COPD: analysis from the TORCH trial. COPD. 2010 Jun;7(3):179-85. doi: 10.3109/15412555.2010.481695. PMID 20486816
- [Background] Marchand E. Effect of pharmacotherapy on rate of decline of FEV(1) in the TORCH study. Am J Respir Crit Care Med. 2009 Mar 1;179(5):426; author reply 426-7. doi: 10.1164/ajrccm.179.5.426. No abstract available. PMID 19234322
- [Background] McGarvey LP, John M, Anderson JA, Zvarich M, Wise RA; TORCH Clinical Endpoint Committee. Ascertainment of cause-specific mortality in COPD: operations of the TORCH Clinical Endpoint Committee. Thorax. 2007 May;62(5):411-5. doi: 10.1136/thx.2006.072348. Epub 2007 Feb 20. PMID 17311843
- [Background] Middleton PG. Management of patients with COPD: a comparison of the INSPIRE and TORCH studies. Am J Respir Crit Care Med. 2008 Jul 1;178(1):106; author reply 106-7. doi: 10.1164/ajrccm.178.1.106. No abstract available. PMID 18565964
- [Background] Miravitlles M, Anzueto A. Insights into interventions in managing COPD patients: lessons from the TORCH and UPLIFT studies. Int J Chron Obstruct Pulmon Dis. 2009;4:185-201. Epub 2009 May 7. PMID 19516917
- [Background] Niewoehner DE. TORCH and UPLIFT: what has been learned from the COPD "mega-trials"? COPD. 2009 Feb;6(1):1-3. doi: 10.1080/15412550902723984. PMID 19229702
- [Background] Calverley PM, Anderson JA, Celli B, Ferguson GT, Jenkins C, Jones PW, Crim C, Willits LR, Yates JC, Vestbo J; TORCH Investigators. Cardiovascular events in patients with COPD: TORCH study results. Thorax. 2010 Aug;65(8):719-25. doi: 10.1136/thx.2010.136077. PMID 20685748
- [Background] Salmeterol plus fluticasone fails to reduce mortality in patients with COPD. Formulary 2007;42:245-6.
- [Background] Stockley RA. Progression of chronic obstructive pulmonary disease: impact of inflammation, comorbidities and therapeutic intervention. Curr Med Res Opin. 2009 May;25(5):1235-45. doi: 10.1185/03007990902868971. PMID 19335322
- [Background] Suissa S, Ernst P, Vandemheen KL, Aaron SD. Methodological issues in therapeutic trials of COPD. Eur Respir J. 2008 May;31(5):927-33. doi: 10.1183/09031936.00098307. Epub 2008 Jan 23. PMID 18216056
- [Background] Vestbo J; TORCH Study Group. The TORCH (towards a revolution in COPD health) survival study protocol. Eur Respir J. 2004 Aug;24(2):206-10. doi: 10.1183/09031936.04.00120603. PMID 15332386
- [Background] Vestbo J, Anderson JA, Calverley PM, Celli B, Ferguson GT, Jenkins C, Knobil K, Willits LR, Yates JC, Jones PW. Adherence to inhaled therapy, mortality and hospital admission in COPD. Thorax. 2009 Nov;64(11):939-43. doi: 10.1136/thx.2009.113662. Epub 2009 Aug 23. PMID 19703830
- [Derived] Paly VF, Naya I, Gunsoy NB, Driessen MT, Risebrough N, Briggs A, Ismaila AS. Long-term cost and utility consequences of short-term clinically important deterioration in patients with chronic obstructive pulmonary disease: results from the TORCH study. Int J Chron Obstruct Pulmon Dis. 2019 May 3;14:939-951. doi: 10.2147/COPD.S188898. eCollection 2019. PMID 31190781
- [Derived] Naya IP, Tombs L, Muellerova H, Compton C, Jones PW. Long-term outcomes following first short-term clinically important deterioration in COPD. Respir Res. 2018 Nov 20;19(1):222. doi: 10.1186/s12931-018-0928-3. PMID 30453972
- [Derived] Jenkins CR, Celli B, Anderson JA, Ferguson GT, Jones PW, Vestbo J, Yates JC, Calverley PM. Seasonality and determinants of moderate and severe COPD exacerbations in the TORCH study. Eur Respir J. 2012 Jan;39(1):38-45. doi: 10.1183/09031936.00194610. Epub 2011 Jul 7. PMID 21737561
- [Derived] Jones PW, Anderson JA, Calverley PM, Celli BR, Ferguson GT, Jenkins C, Yates JC, Vestbo J, Spencer MD; TORCH investigators. Health status in the TORCH study of COPD: treatment efficacy and other determinants of change. Respir Res. 2011 May 31;12(1):71. doi: 10.1186/1465-9921-12-71. PMID 21627828
- [Derived] Celli B, Vestbo J, Jenkins CR, Jones PW, Ferguson GT, Calverley PM, Yates JC, Anderson JA, Willits LR, Wise RA; Investigators of the TORCH Study. Sex differences in mortality and clinical expressions of patients with chronic obstructive pulmonary disease. The TORCH experience. Am J Respir Crit Care Med. 2011 Feb 1;183(3):317-22. doi: 10.1164/rccm.201004-0665OC. Epub 2010 Sep 2. PMID 20813884
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: SCO30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SCO30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SCO30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCO30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SCO30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCO30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCO30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register